CLINICAL TRIAL: NCT05049538
Title: A Pilot Investigation to Determine the Utility of Liquid Biopsies and Tumor Molecular Profiling in Predicting Recurrence in Endometrial Cancer
Brief Title: Determine the Utility of Liquid Biopsies and Tumor Molecular Profiling in Predicting Recurrence in Endometrial Cancers
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA19-0309; NCI-2021-08621 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-09-07; First posted 2021-09-20 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Endometrial Clear Cell Adenocarcinoma; Endometrial Dedifferentiated Carcinoma; Endometrial Mucinous Adenocarcinoma; Endometrial Serous Adenocarcinoma; Malignant Uterine Neoplasm; Uterine Corpus Carcinosarcoma
MeSH Terms: conditions — Uterine Neoplasms | interventions — Liquid Biopsy; Papanicolaou Test; Vaginal Smears

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, Pap smear): Patients undergo collection of blood samples for liquid biopsy during pre-treatment consultation before hysterectomy, after hysterectomy but before starting any chemotherapy, and at the end of last chemotherapy cycle. Patients also undergo collection of tissue samples during hysterectomy. Patients may also undergo Pap smears before and after hysterectomy.
  Interventions: Procedure: Biospecimen Collection; Procedure: Liquid Biopsy; Other: Pap Smear

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples
  Other Names: Biological Sample Collection
Procedure: Liquid Biopsy — Undergo liquid biopsy
  Other Names: Plasma Biopsy
Other: Pap Smear — Undergo Pap smear
  Other Names: Cervical Smear Preparation; Cervical Smear Procedure; Pap Smear Procedure; Pap Test; Papanicolaou Smear Procedure; Papanicolaou Test; Vaginal Smears

SUMMARY:
This study is to find out how well liquid biopsies work as a non-invasive alternative to other methods of finding cancer cells (such as a tissue biopsy) in patients with endometrial cancer. A liquid biopsy is a blood test that may be able to find cancer cells. Collecting and storing samples of blood and tissue from patients with endometrial cancer to study in the laboratory may help doctors learn how the cells in the blood may change during treatment for uterine cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare TP53, FBXW7, and other mutated gene variant allele frequencies (VAF) in serial circulating cell free deoxyribonucleic acid (ccfDNA) samples obtained from patients with endometrial cancer subtypes during the primary treatment course, which may include pretreatment, post-surgical removal, post adjuvant treatment, and at time of recurrence.

II. Compare the findings from the liquid biopsy mutational analysis to next generation sequencing from the primary tumor.

EXPLORATORY OBJECTIVES:

I. To estimate the presence of malignant cells in the vagina before and after minimally invasive hysterectomy among patients with endometrial cancer.

II. Characterize the immune profile and single cell ribonucleic acid (RNA) sequencing (scRNAseq) profile of endometrial cancer subtypes.

III. Estimate time to progression (TTP), and investigate potential correlations between mutated gene variant allele frequency (VAF) ccfDNA samples and progression.

IV. Compare the efficacy of experimental ccfDNA assays to approved ccfDNA assay using the same samples.

OUTLINE:

Patients undergo collection of blood samples for liquid biopsy during pre-treatment consultation before hysterectomy, after hysterectomy but before starting any chemotherapy, and at the end of last chemotherapy cycle. Patients also undergo collection of tissue samples during hysterectomy. Patients may also undergo Pap smears before and after hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 years and older
* Histologic diagnosis of endometrial cancer
* Candidate for primary surgical treatment or has recently had prior primary surgery
* Willing and able to provide informed consent

Exclusion Criteria:

Patients who have received prior treatment including chemotherapy or radiation therapy for endometrial cancer. Patients with prior primary surgery will be allowed to enroll in this trial if the patient has not received any chemotherapy or radiation at the time of enrollment. Note: patients with a history of other cancers may be enrolled after discussion with the PI if it is determined that they are at low risk for recurrence or metastasis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of uterine cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of circulating cell free deoxyribonucleic acid (ccfDNA) mutations | through study completion, an average of 1 year
  The proportion of ccfDNA mutations determined by liquid biopsy will be calculated along with 95% confidence intervals, and comparison between treatment time points will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela T Soliman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org